CLINICAL TRIAL: NCT06894225
Title: Proof-of-Concept Study of ACT001 in Adult Patients With Recurrent Glioblastoma Harbouring STAT3-High Signature
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Neuroscience Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-3595
Record Dates: First submitted 2024-11-27; First posted 2025-03-25 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Recurrent Glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — ACT001

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- ACT001 (Experimental)
  Interventions: Drug: ACT001

INTERVENTIONS:
Drug: ACT001 — Patients recruited and have signed informed consent will be initiated on ACT001 400mg twice a day. Treatment course will repeat every 28 days in the absence of disease progression or unacceptable toxicity

SUMMARY:
This trial will study the effectiveness of ACT001 in adult patients whose Glioblastoma have recurred with a STAT3-high signature after standard-of-care treatment with at least radiation therapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of GBM according to 2021 WHO classification
* Availability of tumor tissue representative of GBM from definitive surgery or biopsy and tested to harbour STAT3-High Signature
* Previous treatment with at least radiation therapy
* Documented recurrence of malignant glioma by diagnostic biopsy, resection or MRI performed within 21 days of study enrolment per RANO criteria.

There is no limit on number of previous recurrences or lines of treatment

* At least 12 weeks after the end of prior radiation therapy is required unless there is either: i) histopathologic confirmation of recurrent tumor, or ii) n new enhancement on MRI outside of the radiation treatment field
* An interval of at least 4 weeks after the last administration of any investigational agent or any other treatment prior to first dose of STAT3 inhibitor
* Age 21 years or older on the day of signing informed consent
* Karnofsky performance status (KPS) of 70 or higher
* Patient has adequate bone marrow, renal, and hepatic function ≤ 21 days prior to study enrolment (Step 2) as follows:

  * Absolute neutrophil count (ANC) ≥1,500/mm3
  * Platelets ≥ 100,000/mm3
  * Hemoglobin (Hgb) ≥ 9.0 g/dL (Note: The use of transfusion or other intervention to achieve Hgb ≥ 9.0 g/dL is acceptable.)
  * Renal function: calculated creatinine clearance ≥ 30 mL/min by the Cockcroft-Gault formula
  * Hepatic function: Total bilirubin, Aspartate Aminotransferase (AST), and Alanine Aminotransferase (ALT) ≤ 1.5 times upper limit of normal (ULN). Patients with Gilbert's syndrome documented in medical history may be enrolled if bilirubin is < 3 times ULN.

Exclusion Criteria:

* Presence of extracranial metastatic or leptomeningeal disease
* Previous or current treatment with a JAK or STAT3 inhibitor
* Previous or current treatment with bevacizumab/VEGF inhibitor
* Patient is a lactating or pregnant female.
* Symptomatic intra-tumoural haemorrhage
* Severe, active co-morbidity, defined as follows:

  * Patients with clinically defined Acquired Immune-Deficiency Syndrome (AIDS)-defining illness.
  * Active connective tissue disorders, such as lupus or scleroderma, that in the opinion of the Investigator may put the patient at high risk of toxicity
  * Any other major medical illnesses or psychiatric impairments that in the Investigator's opinion will prevent administration or completion of protocol therapy

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate | 1.5 years
  ORR as defined as radiographic complete response, or partial response, or stable disease. Patients with stable disease will be considered responders if disease is stable for 24 weeks or more. The regimen will be considered worthy of further study if responses as defined above are observed in at least 3 of the 12 patients.

SECONDARY OUTCOMES:
Progression-free survival (PFS) & Overall survival (OS) | 1.5 years
  6 months progression-free survival (PFS), defined as proportion of patients who remained alive and progression-free at 6 months.
  PFS, which is defined as time from study enrolment to progression of disease per RANO criteria, or death, whichever occurs first. For patients who are not documented to have experienced a PFS event at the time of an analysis, PFS will be right-censored on the date of their last adequate assessment of disease.
  Overall survival (OS), which is defined as time from study enrolment to death from any cause. For patients who are not reported to have died at the time of an analysis, OS will be right-censored at the last date the patient is documented to be alive.

OTHER OUTCOMES:
Toxicity evaluation | 1.5 years
  Study team will assess adverse events, laboratory data and vital signs throughout the study. Analyses of adverse events will include only "treatment-emergent" events, i.e., those that start or worsen on or after the day of the first dose of study drug. Adverse event severity and laboratory evaluation changes will be assessed by utilizing National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0. Adverse events will be summarized by preferred terms within a System and Organ Class according to the most current Medical Dictionary for Regulatory Activities (MedDRA) dictionary. Changes from baseline will be analyzed for each scheduled post-baseline visit and for the final visit for blood chemistry and hematology parameters, as well as urinalysis and vital sign parameters. Shifts in laboratory values from baseline NCI CTCAE grades to maximum and final post-baseline grades will be assessed.
Drug levels | 1.5 years
  Drug levels in cerebrospinal fluid and tissue sample when available in patients who are agreeable to proceed with Omaya shunt insertion, lumbar puncture or undergoes further surgical resection following treatment with ACT001.
Treatment response and resistance | 1.5 years
  Tissue and blood exosome biomarkers that are predictive of treatment response and treatment resistance.

CONTACTS AND LOCATIONS:
Locations (1):
- National Neuroscience Institute, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No